CLINICAL TRIAL: NCT06532760
Title: Identification Des Fragments de Canaux Sodiques Comme Biomarqueurs sériques d'Une lésion Traumatique du système Nerveux Central
Brief Title: Identification of Sodium Channel Fragments as Serum Biomarkers of a Traumatic Central Nervous System Injury
Acronym: SpasT-SCI-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM21_0427
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injury; Spasticity, Muscle; Brain Injuries
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity; Brain Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 3 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Spinal cord injury (Experimental)
  Interventions: Other: Blood sampling
- Patients with Brain Injury (Active Comparator)
  Interventions: Other: Blood sampling
- Healthy volunteers (Active Comparator)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling to study sodium fragment kinetics

SUMMARY:
Following spinal cord injury (SCI), 75% of patients develop spasticity of the limbs characterized by an increase in muscle tone causing severe pain. Currently, the diagnosis of spinal cord injury is based on clinical and radiological evaluation by CT and MRI, but there is no reliable biomarker capable of predicting the medium and long-term clinical course in terms of emergence and severity of spasticity and neurological recovery. Recently, pre-clinical models in rats have shown the presence of protein fragments from a cleavage of sodium channels in spinal cords below the level of injury. Other studies have also shown the presence of these fragments in the brain following a head injury. These fragments would be potentially useful as a biomarker of the SCI. The detection of sodium fragments would be potentially useful as a biomarker of a lesion of the central nervous system (spinal cord or brain) and of the severity of the spasticity in patients suffering from SCI. The main objective of this study is to detect the presence of sodium fragments in blood samples from patients with SCI from or brain injury. The secondary objectives will be to study the post-lesional / injury kinetics of sodium fragments, to determine their diagnostic values in terms of the severity of the injury, and their prognostic values concerning the emergence of the spasticity in patients with SCI. An initial prospective cohort will include 40 people. The fragments of sodium channels will be measured in blood samples taken within 6 hours post-trauma, then 1, 3, 5 and 7 days post-trauma, as well as 3 and 6 months post-trauma. The overall expression of sodium fragments will be compared to that of healthy controls. Participants will be recruited in the acute care units of the AP-HM. Participants will be recruited from the main acute care units of the AP-HM. Post-traumatic follow-up assessments during their rehabilitation will be carried out at 3 and 6 months in the neurosurgery department of North Hospital from APHM.

ELIGIBILITY:
healthy volonteers group: Inclusion Criteria

* Male or Female
* Age 18 to 75
* free of central or peripheral nervous system trauma
* Having given free and informed consent
* Beneficiary of or affiliated to a social security scheme

Exclusion Criteria:

* Pregnant or breast-feeding women
* Person under guardianship or curatorship
* Diagnosis of a neurological disorder
* Diagnosis of a psychiatric disorder
* Diagnosis of a neurodegenerative disease

Spinal Cord injury patients group:

Inclusion Criteria:- Male or female

* Aged 18 to 75
* Beneficiary of or affiliated to a social security scheme
* Having suffered within 6 hours a trauma with an acute LME confirmed according to the following characteristics:
* Lesion located at C4-T12 level and radiologically documented (CT scan and/or spinal MRI performed within 6 hours)
* Complete or incomplete according to the American Spinal Injury Association impairment scale (ASIA A to D)
* Signed consent for emergency and continuation of study

Exclusion criteria:

* Pregnant or breast-feeding patient
* Absence of consent from the volunteer or his/her trusted support person
* Patient under guardianship or trusteeship
* Brain injury due to cranioencephalic trauma with a Glasgow score of less than 14 on reassessment, associated with a cerebral CT scan of grade III or less on the Marshall classification
* Presence of another neurological or mental disorder or neurodegenerative disease

Brain injury patients Group:

Inclusion criteria:

* Male or female
* Aged 18 to 75
* Have suffered a traumatic brain injury (TBI) with a proven acute brain injury according to the following characteristics:
* Glasgow score less than 13 on admission without metabolic cause in the context of head trauma
* Cerebral CT scan at least grade II according to Marshall classification
* Absence of traumatic spinal lesion threatening the integrity of the spinal canal assessed by neuroradiological examination (CT and/or MRI)
* Signed consent for emergency and continuation of study
* ASIA E score

Exclusion criteria:

* Pregnant or breast-feeding patient
* Absence of consent from the volunteer or his/her trusted support person
* Patient under guardianship
* ASIA score A to D
* Presence of another neurological or mental disorder or neurodegenerative disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Detect the presence of sodium fragments in blood samples from patients | 6 hours to 6 months post-injury

SECONDARY OUTCOMES:
kinetics of sodium fragments in patients with acute SCI and in traumatic brain injury patients in the post-trauma period | 6 hours to 6 months post-injury
To correlate measurements of sodium fragments in blood from 6 hours to 6 months post-injury with the occurence of spasticity in the post-trauma period | 3 and 6 months-post-injury

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — francois.cremieux@ap-hm.fr

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baucher G, Liabeuf S, Brocard C, Ponz A, Baumstarck K, Troude L, Leone M, Roche PH, Brocard F. The SpasT-SCI-T trial protocol: Investigating calpain-mediated sodium channel fragments as biomarkers for traumatic CNS injuries and spasticity prediction. PLoS One. 2025 May 21;20(5):e0319635. doi: 10.1371/journal.pone.0319635. eCollection 2025. PMID 40397864